CLINICAL TRIAL: NCT00075335
Title: Peripheral Blood Hematopoietic Progenitor Cell Mobilization With AMD 3100 (Mozobil) in Healthy Volunteers Previously Mobilized With G-CSF
Brief Title: AMD 3100 (Mozobil Plerixafor) to Mobilize Stem Cells for Donation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Richard Childs, M.D., Hematology Clinician, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040078; 04-H-0078 (Other: NIH NHLBI)
Record Dates: First submitted 2004-01-08; First posted 2004-01-09 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: Hematopoietic Stem Cells; Mobilization; Alloreactivity; T Cell Polarization; Dendritic Cells; Plerixafor; Mozobil; Healthy Volunteer (HV)
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMD 3100 (Mozobil plerixafor) (Experimental): AMD 3100 (Mozobil plerixafor)mobilized peripheral blood hematopoietic progenitor cells from healthy volunteers will be characterized by cellular content and immunological properties.
  Interventions: Drug: AMD3100 (Mozobil plerixafor)

INTERVENTIONS:
Drug: AMD3100 (Mozobil plerixafor) — AMD 3100 (Mozobil plerixafor)mobilized peripheral blood hematopoietic progenitor cells from healthy volunteers will be characterized by cellular content and immunological properties.
  Other Names: Mozobil plerixafor

SUMMARY:
Peripheral blood progenitor cells (PBPC) have become the preferred source of hematopoetic stem cells for allogeneic transplantation because of technical ease of collection and shorter time required for engraftment. Traditionally, granulocyte-colony stimulating factor (G-CSF) has been used to procure the peripheral blood stem cell graft. Although regimens using G-CSF usually succeed in collecting adequate numbers of PBPC from healthy donors, 5%-10% will mobilize stem cells poorly and may require multiple large volume apheresis or bone marrow harvesting. Although G-CSF is generally well tolerated in healthy donors, it may be associated with bone pain, headache, myalgia and rarely life threatening side effects like stroke, myocardial infarction and splenic rupture.

AMD3100, is a bicyclam compound that inhibits the binding of stromal cell derived factor-1 (SDF-1) to its cognate receptor CXC- chemokine receptor 4 (CXCR4). CXCR4 is present on cluster of differentiation 34 (CD34)+ hematopoetic progenitor cells and its interaction with stromal cell derived factor 1 (SDF-1) plays a pivotal role in the homing of CD34+ cells in the bone marrow. Inhibition of the CXCR4-SDF1 axis by AMD3100 releases CD34+ cells into the circulation, which can then be collected easily by apheresis.

Recently, a published report demonstrated that large numbers of CD34+ cells were rapidly mobilized in healthy volunteers following a single subcutaneous injection of AMD3100. Remarkably, the number of CD34+ cells collected by apheresis following a single injection of AMD3100 was comparable to the number of CD34+ cells collected from historical controls receiving 5 days of G-CSF prior to stem cell mobilization.

In this study we will collect PBPCs following a single subcutaneous injection of AMD3100 from healthy donors who have previously had PBPC collected using standard G-CSF mobilization. The AMD3100 mobilized cells, G-CSF mobilized cells, and circulating cells prior to both AMD3100 and G-CSF mobilization will be analyzed in terms of cellular content and function of lymphocytes, natural killer (NK) cells, and antigen presenting cells. AMD3100 mobilized PBPC will be collected for the purpose of research studies and will not be used for therapeutic purposes.

DETAILED DESCRIPTION:
Peripheral blood progenitor cells (PBPC) have become the preferred source of hematopoietic stem cells for allogeneic transplantation because of technical ease of collection and shorter time required for engraftment. Traditionally, granulocyte-colony stimulating factor (G-CSF) has been used to procure the peripheral blood stem cell graft. Although regimens using G-CSF usually succeed in collecting adequate numbers of PBPC from healthy donors, 5%-10% will mobilize stem cells poorly and may require multiple large volume apheresis or bone marrow harvesting. Although G-CSF is generally well tolerated in healthy donors, it may be associated with bone pain, headache, myalgia and rarely life threatening side effects like stroke, myocardial infarction and splenic rupture.

AMD3100 is a bicyclam compound that inhibits the binding of stromal cell derived factor-1 (SDF-1) to its cognate receptor CXCR4. CXCR4 is present on CD34+ hematopoietic progenitor cells and its interaction with SDF-1 plays a pivotal role in the homing of CD34+ cells in the bone marrow. Inhibition of the CXCR4-SDF1 axis by AMD3100 releases CD34+ cells into the circulation, which can then be collected easily by apheresis. Recently, a published report demonstrated that large numbers of CD34+ cells were rapidly mobilized in healthy volunteers following a single subcutaneous injection of AMD3100. Remarkably, the number of CD34+ cells collected by apheresis following a single injection of AMD3100 was comparable to the number of CD34+ cells collected from historical controls receiving 5 days of G-CSF prior to stem cell mobilization. Although the study population is relatively small, side-effects to this agent have been mild and transient with no serious complications having been reported. The ability to collect a large quantity of PBPC with a single injection of this drug makes this an attractive agent for mobilizing donors of allogeneic PBPC. However, the immunologic profiles of AMD3100 mobilized cells, in terms of lymphocyte content (T cell, B cell, NK cell, immuno-regulatory T cell), T cell polarization status (TH1 versus TH2), status of antigen presenting cells (DC1 versus DC2), alloreactive potential, and preservation of reactivity to infectious agents [e.g. Epstein Barr Virus (EBV), Cytomegalovirus (CMV)] are unknown. Consequently, whether AMD3100 mobilized PBPC would be suitable for use as an allograft is uncertain. In this study we will collect PBPCs following a single subcutaneous injection of AMD3100 from healthy donors who have previously had PBPC collected using standard G-CSF mobilization. The AMD3100 mobilized cells, G-CSF mobilized cells, and circulating cells prior to both AMD3100 and G-CSF mobilization will be analyzed in terms of cellular content and function of lymphocytes, NK cells, and antigen presenting cells. AMD3100 mobilized PBPC will be collected for the purpose of research studies and will not be used for therapeutic purposes.

The primary objective is to characterize the immunological properties of AMD3100 mobilized (cytokine gene expression profiles) T-cells compared to G-CSF mobilized T-cells.

Secondary endpoints include the cellular content and other immune properties of AMD3100 mobilized cells yields of hematopoietic progenitor cells, immune cells, and other cellular subsets collected by apheresis in subjects undergoing G-CSF and AMD3100 mobilization and the safety profile of AMD3100.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Mobilization and collection of PBPC using G-CSF at least 60 days prior to protocol enrollment (stem cell donors enrolled on Branch transplant protocols or healthy volunteers enrolled on 96-H-0049: Use of granulocyte colony stimulating factor mobilized leukapheresis collections from healthy volunteers).
  2. Ages greater than or equal to 18 years and less than or equal to 80 years.
  3. Normal renal function: creatinine less than 1.5 mg/dl.
  4. Normal liver function: total bilirubin less than 1.5mg/dl, alanine aminotransferase (ALT) 6 -41 U/L, aspartate aminotransferase (AST) 9-34 U/L.
  5. Normal blood count: white blood cell (WBC) 3000-10000/mm(3)

     granulocytes greater than 1500/mm(3)

     platelets greater than 150,000/mm(3)

     hemoglobin (females greater than 11.1 g/dl, males greater than 12.7 g/dl).
  6. Subject must be eligible for normal blood donation and fit to undergo apheresis procedure (antecubital veins must be adequate for peripheral access during apheresis).
  7. Ability to comprehend the investigational nature of the study and provide informed consent.

EXCLUSION CRITERIA: Any of the Following

1. Active infection or history of recurrent infection- hepatitis B and C (HBsAg, Anti-HBc, Anti-HCV), HIV and human T- lymphocytic virus (HTLV-1).
2. History of autoimmune disease such as rheumatoid arthritis, systemic lupus erythematous.
3. History of cancer within the past 5 years excluding basal cell or squamous cell carcinoma of the skin.
4. History of any hematologic disorders including thromboembolic disease.
5. History of cardiac disease such as uncontrolled hypertension, peripheral vascular disease, myocardial infarction, cardiac arrhythmias OR related symptoms such as tachycardia, chest pain, shortness of breath which have required medical intervention OR treatment or a Framingham coronary disease risk prediction score of greater than 10% 10 year coronary heart disease (CHD) risk.
6. History of cerebrovascular disease, transient ischemic attack, or stroke.
7. Pregnant or lactating.
8. Severe psychiatric illness: mental deficiency sufficiently severe as to make informed consent impossible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mohle R, Murea S, Kirsch M, Haas R. Differential expression of L-selectin, VLA-4, and LFA-1 on CD34+ progenitor cells from bone marrow and peripheral blood during G-CSF-enhanced recovery. Exp Hematol. 1995 Dec;23(14):1535-42. PMID 8542944
- [Background] Mohle R, Haas R, Hunstein W. Expression of adhesion molecules and c-kit on CD34+ hematopoietic progenitor cells: comparison of cytokine-mobilized blood stem cells with normal bone marrow and peripheral blood. J Hematother. 1993 Winter;2(4):483-9. doi: 10.1089/scd.1.1993.2.483. PMID 7522108
- [Background] Petit I, Szyper-Kravitz M, Nagler A, Lahav M, Peled A, Habler L, Ponomaryov T, Taichman RS, Arenzana-Seisdedos F, Fujii N, Sandbank J, Zipori D, Lapidot T. G-CSF induces stem cell mobilization by decreasing bone marrow SDF-1 and up-regulating CXCR4. Nat Immunol. 2002 Jul;3(7):687-94. doi: 10.1038/ni813. Epub 2002 Jun 17. PMID 12068293
- [Result] Lundqvist A, Smith AL, Takahashi Y, Wong S, Bahceci E, Cook L, Ramos C, Tawab A, McCoy JP Jr, Read EJ, Khuu HM, Bolan CD, Joo J, Geller N, Leitman SF, Calandra G, Dunbar C, Kurlander R, Childs RW. Differences in the phenotype, cytokine gene expression profiles, and in vivo alloreactivity of T cells mobilized with plerixafor compared with G-CSF. J Immunol. 2013 Dec 15;191(12):6241-9. doi: 10.4049/jimmunol.1301148. Epub 2013 Nov 15. PMID 24244025
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-H-0078.html

RESULTS

PARTICIPANT FLOW:
Groups:
- AMD 3100 (Mozobil Plerixafor ) Volunteers: Peripheral blood hematopoietic progenitor cell mobilization with AMD 3100 (Mozobil plerixafor) in healthy volunteers. AMD 3100 volunteer response to peripheral blood stem cell mobilization
Period: Overall Study
Arm/Group | AMD 3100 (Mozobil Plerixafor ) Volunteers
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AMD 3100 (Mozobil Plerixafor ) Volunteers: Peripheral blood hematopoietic progenitor cell mobilization with AMD 3100 (Mozobil plerixafor) in healthy volunteers
Arm/Group | AMD 3100 (Mozobil Plerixafor ) Volunteers
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Cytokine Gene Expression Profiles (84 Genes) in T Cells Following G-CSF Administration
Description: Examine G-CSF mobilization effect on cytokine polarization of T-cells. Analyze cytokine gene expression profiles using a Th1-Th2-Th3 RT-PCR plate in CD3+ T cells collected form subjects mobilized with 5 injections of G-CSF. 84 cytokine genes were analyzed for significant alteration in their profiles.
Time Frame: 1 Day
Population: 8 Subjects received G-CSF for 5 days.
Measure: Number; unit: unique cytokine genes affected
Groups:
- AMD 3100 Volunteers: Peripheral blood hematopoietic progenitor cell mobilization with AMD 3100 (Mozobil plerixafor) in healthy volunteers
Arm/Group | AMD 3100 Volunteers
Number analyzed (Participants) | 8
unique cytokine genes affected | 16

2. Primary Outcome: Change in Cytokine Gene Expression Profiles (84 Genes) in T Cells Following Plerixafor Administration
Description: Examine plerixafor mobilization effect on cytokine polarization of T-cells. Analyze cytokine gene expression profiles using a Th1-Th2-Th3 RT-PCR plate in CD3+ T cells collected form subjects mobilized with a single injection of plerixafor. 84 cytokine genes were analyzed for significant alteration in their profiles.
Time Frame: 1 Day
Population: Subjects who received plexirxafor 240mcg/kg. Data was collected 6 hours after injection.
Measure: Number; unit: unique cytokine genes affected
Arm/Group | AMD 3100 Volunteers
Number analyzed (Participants) | 8
unique cytokine genes affected | 0

ADVERSE EVENTS:
Arm/Group | AMD 3100 (Mozobil Plerixafor ) Volunteers
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMD 3100 (Mozobil Plerixafor ) Volunteers (N=8)
elevated LDH (Blood and lymphatic system disorders) | 1
elevated Lymphs (efficacy measure) (Blood and lymphatic system disorders) | 7
elevated lymphs (expected) (Blood and lymphatic system disorders) | 1
elevated Monos (expected) (Blood and lymphatic system disorders) | 8
elevated Polys (expected) (Blood and lymphatic system disorders) | 8
elevated WBCs (expected) (Blood and lymphatic system disorders) | 8
Sinus tachycardia (rate 103) (Cardiac disorders) | 1
auditory (R ear) pain (Ear and labyrinth disorders) | 1
Cramps, abdominal (Gastrointestinal disorders) | 1
feel need to vomit, no nausea (Gastrointestinal disorders) | 1
Headache (General disorders) | 2
Hot feeling (General disorders) | 1
Swelling, leg (General disorders) | 1
Injection site (erythema) (Immune system disorders) | 5
Injection site (induration) (Immune system disorders) | 2
Injection site (pain) (Immune system disorders) | 3
Injection site (pruritus) (Immune system disorders) | 1
muscle pain (Musculoskeletal and connective tissue disorders) | 1
paresthesia (facial tingling) (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No